CLINICAL TRIAL: NCT06135350
Title: A Randomized, Double-blind, Placebo Controlled Clinical Trial to Study the Efficacy and Safety of the Drug Fluorothiazinone (Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation) in Prophylaxis of Nosocomial Bacterial Infections With Participation of Patients on Mechanical Ventilation
Brief Title: Clinical Trial to Study the Efficacy and Safety of Fluorothiazinone (N.F. Gamaleya NRCEM) in Prophylaxis of Nosocomial Bacterial Infections With Participation of Patients on MV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 06-FT-2021, v. 3.0, 03.11.2022
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-05

CONDITIONS: Gram Negative Pneumonia; Gram-Negative Bacterial Infections; Bacteremia Caused by Gram-Negative Bacteria
MeSH Terms: conditions — Gram-Negative Bacterial Infections | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental)
  Interventions: Drug: Fluorothiazinone, tablets 300 mg at a dose of 2400 mg/day
- Placebo arm (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fluorothiazinone, tablets 300 mg at a dose of 2400 mg/day — Treatment arm patients will receive Fluorothiazinone, tablets 300 mg at a dose:
  * 2400 mg/day (4 tablets twice a day) for the first 2 days and;
  * 1800 mg/day (3 tablets twice a day) from the third day and further (but no more than 14 days) until the occurrence of ventilator-associated pneumonia caused by gram-negative bacteria, confirmed clinically and microbiologically, OR the completion of the patient's participation in the study for other reasons.
  Tablets are taken 2 times a day 12 hours apart 30 minutes after meal, no more than 14 days.
  Arms: Treatment arm
Other: Placebo — Placebo arm patients will receive placebo:
  * 4 tablets twice a day for the first 2 days and;
  * 3 tablets twice a day and further (but no more than 14 days) until the occurrence of ventilator-associated pneumonia caused by gram-negative bacteria, confirmed clinically and microbiologically, OR the completion of the patient's participation in the study for other reasons.
  Tablets are taken 2 times a day 12 hours apart 30 minutes after meal, no more than 14 days.
  Arms: Placebo arm

SUMMARY:
This study is designed to evaluate the clinical and antibacterial efficacy, safety and pharmacokinetics of the drug Fluorothiazinone compared to placebo to prevent nosocomial gram-negative bacterial infections with participation of patients on mechanical ventilation.

The main objectives of this study are:

* Evaluation of the clinical and antibacterial efficacy of the drug Fluorothiazinone in combination with standard measures for the prevention of nosocomial infections compared to placebo in combination with standard measures for the prevention of nosocomial infections for the prevention of nosocomial infections caused by bacterial gram-negative flora in patients on mechanical ventilation.
* Evaluation of the safety and tolerability of the drug Fluorothiazinone in patients on mechanical ventilation.
* Evaluation of the pharmacokinetics (in whole blood) of the drug Fluorothiazinone with a single daily dose of 2400 mg/day.

Researchers will compare results for the treatment and the placebo arms.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's written consent to participate in the study in accordance with the current legislation or the decision of the board in case of absence of consciousness of the patient.
2. Patients are at least 18 years old, male and female.
3. Patients who are in the ICU (intensive care unit).
4. Patients with:

   4.1. Laboratory confirmed SARS-CoV-2 (Severe acute respiratory syndrome-related coronavirus-2) on screening (a patient's coronavirus infection can be confirmed either before admission to the hospital (for outpatient treatment) or when admitted to the hospital) by RT-PCR (reverse transcription polymerase chain reaction) AND severe community-acquired pneumonia in ICU with evidence of viral lung injury and symptoms of respiratory failure:
   * SpO2 (peripheral oxygen saturation) ≤ 93%;
   * Lung changes of 3rd- to 4th-degree according to CT (results of computed tomography), consistent with viral involvement; OR 4.2. Acute stroke; OR 4.3. Acute heart failure: Cardiogenic shock of any cause, pulmonary edema, or acute decompensated chronic heart failure.
5. Patients who have been on ALV (artificial lung ventilation) for no more than 12 hours.
6. Patients who are according to the investigator are at high risk to be transferred to ALV within 72 hours of the initiation of the therapy.
7. All women of childbearing age and men with partners of childbearing age should agree to use an effective contraceptive methods (e.g., implants, infections, combination oral contraceptives, intrauterine device, abstinence, vasectomy or vasectomy partner) during the entire study.

Exclusion Criteria:

1. The patient was not switched to ALV within 72 hours (3 days) after receiving the investigational drug.
2. People who have a bloodstream infection, identified during the screening.
3. A patient may terminate his/her participation in the study at any time for any reason and without any explanation.

3. The investigator may also decide to terminate the patient's participation at any time if it is required due to the patient's condition.

4. The sponsor or the regulator may also request the trial to be terminated early, either due to how the trial was conducted, or due to application safety data, or other reasons.

5. The main reasons why the patient may withdraw from the study are:

* Refusal of the patient to participate in the study;
* Development of an AE (adverse event) / SAE (serious adverse event) that prevents further study participation;
* The occurrence of concomitant somatic diseases / symptoms or exacerbation of chronic diseases not related to the investigational drug (at the discretion of the medical investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MV-associated pneumonia caused by gram-negative bacteria (72-120 hours from the moment of tracheal intubation and the start of the MV) | Throughout the therapy period (14 days).
  The proportion of patients in the study groups without clinically and microbiologically confirmed MV-associated pneumonia caused by gram-negative bacteria, which developed no earlier than 72 hours (3 days) and no later than 120 hours (5 days) from the moment of tracheal intubation and the start of the MV, in the absence of signs of pulmonary infection at the time of intubation.

SECONDARY OUTCOMES:
Time from the beginning of the MV to the development of MV-associated pneumonia | Throughout the therapy period (14 days).
  The time from the beginning of the MV to the development of MV-associated pneumonia caused by gram-negative bacteria, confirmed clinically and microbiologically, in the study groups during the entire period of therapy.
Time from the beginning of the MV to the development of a bloodstream infection | Throughout the therapy period (14 days).
  The time from the beginning of the MV to the development of a bloodstream infection caused by gram-negative bacteria, confirmed microbiologically in the study groups during the entire period of therapy.
Time from the beginning of the MV to the development of urinary tract infection | Throughout the therapy period (14 days).
  The time from the beginning of the MV to the development of urinary tract infection caused by gram-negative bacteria, confirmed microbiologically in the study groups during the entire period of therapy.
Proportion of patients who developed urinary tract infection | Throughout the therapy period (14 days).
  The proportion of patients who developed urinary tract infection caused by gram-negative bacteria, confirmed microbiologically, in the study groups during the entire period of reception of the investigative drug (IMP).
Proportion of patients who did not develop MV-associated pneumonia | Throughout the therapy period (14 days).
  The proportion of patients who did not develop MV-associated pneumonia caused by gram-negative bacteria, confirmed clinically and microbiologically, in the study groups during the entire period of reception of the investigative drug (IMP).
Proportion of patients who have gram-negative bacteria | Throughout the therapy period (14 days).
  The proportion of patients who have gram-negative bacteria isolated from the respiratory tract, with no clinical picture of pneumonia.
Proportion of patients who developed a bloodstream infection (during the entire period of therapy) | Throughout the therapy period (14 days).
  The proportion of patients who developed a bloodstream infection caused by gram-negative microflora, confirmed microbiologically in the study groups during the entire period of therapy.
Proportion of patients who developed a bloodstream infection (after the patient was transferred to the MV) | Throughout the therapy period (14 days).
  The proportion of patients who developed a bloodstream infection caused by gram-negative microflora, confirmed microbiologically in the study groups after the patient was transferred to the MV.
Proportion of patients with septic complications | Throughout the therapy period (14 days).
  The proportion of patients with septic complications in the study groups during the entire period of therapy.
The proportion of fatal outcomes | Throughout the therapy period (14 days).
  The proportion of fatal outcomes in the study groups during the entire period of therapy.

OTHER OUTCOMES:
Comparative characteristics of colonization of the respiratory and urinary tracts | Throughout the therapy period (14 days).
  Comparative characteristics of colonization of the respiratory and urinary tracts by individual pathogens in patients on the MV.
Comparative assessment of the condition on the SOFA scale | Throughout the therapy period (14 days).
  Comparative assessment of the condition on the Sequential Organ Failure Assessment (SOFA) scale. Comparative assessment of the condition on the SOFA scale throughout the study. Score ranges from 0 (best) to 24 (worst) points.
Comparative assessment of the condition on the APACHE II scale | Throughout the therapy period (14 days).
  Comparative assessment of the condition on the Acute Physiology and Chronic Health Evaluation II (APACHE II) scale throughout the study. Calculates an integer score from 0 to 71 based on multiple measurements. Higher scores correspond to more severe disease and a higher risk of death.

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - State Budgetary Healthcare Institution of Moscow City Clinical Hospital No. 1 named after N.I. Pirogov of the Moscow Department of Health (State Clinical Hospital No. 1 named after N.I. Pirogov), Moscow, Moscow
  - City Clinical Hospital No. 24 of the Moscow City Department of Health, Moscow, Moscow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://grls.minzdrav.gov.ru/CIPermissionMini.aspx?CIStatementGUID=5281d32d-b391-401d-b48a-123aff27f55f&CIPermGUID=f29a6b9f-2c24-426c-94fb-0275d300f2ee